CLINICAL TRIAL: NCT04946916
Title: Validation of Serum Neurofilament Light Chain as a Biomarker to Differentiate Cognitive Impairment From Neurodegenerative or Psychiatric Diseases
Brief Title: Neurofilament Light Chains and Cognitive Impairment in Chronic Psychiatric Disease
Acronym: Nfl_COG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A00695-34
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Bipolar Disorder; Alzheimer Disease; FTD
Keywords: dementia; biomarker
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Four groups of participants will be recruited: participant with psychiatric condition without cognitive impairment, participants with psychiatric condition with cognitive impairment, participants with biological Alzheimer's disease, and participant with fronto-temporal dementia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participant with psychiatric condition without cognitive impairment (Experimental): In the psychiatric condition group without cognitive impairment will be included participants with schizophrenia or bipolar disorder according to DSM V criteria.
  Interventions: Diagnostic Test: blood sample taken
- Participant with psychiatric condition with cognitive impairment (Experimental): In the psychiatric condition group with cognitive impairment will be included participants with schizophrenia or bipolar disorder according to DSM V criteria. To date, there are no clinical criteria for defining the dementia evolution of psychiatric disorders. The diagnosis of psychiatric disorder with cognitive involution is often made on the basis of subjective criteria or on the appreciation of health care teams. In the present study, cognitive involution will be defined by the occurrence of cognitive deterioration objectified by disturbed neuropsychological tests and the occurrence of progressive behavioral changes contrasting with the person's previous state and reported by the care team, a member of the family or by the patient himself. Cognitive involution must be accompanied by a decrease in autonomy with respect to the person's previous abilities.
  Interventions: Diagnostic Test: blood sample taken
- Patients with biological Alzheimer's disease (Experimental): Alzheimer's disease with frontal, amnestic, language, and visual presentation with typical Alzheimer CSF according to the 2011 NIA-AA diagnostic criteria.
  Interventions: Diagnostic Test: blood sample taken
- Patient with fronto-temporal dementia (Experimental): Probable or definite Fronto-temporal dementia, mostly behavioral variant of FTD (according to the diagnostic criteria for FTDb of Rascovsky, 2011) but Semantic Disease, Primary Progressive Non-Fluent Aphasia, Progressive Supra-Nuclear Palsy-DFT will be accepted if behavioral onset.
  Interventions: Diagnostic Test: blood sample taken

INTERVENTIONS:
Diagnostic Test: blood sample taken — Comparaison of Neurofilament light chain serum concentration between the arms
  Other Names: Cognitive tests and psychiatric questionnaires

SUMMARY:
The validation of biomarkers allowing the discrimination of cognitive and behavioral disorders of psychiatric origin from those of neurodegenerative origin would facilitate diagnosis and improve patient management. Neurofilaments, which are markers of neuronal lysis, appear to be a promising biomarker. In a previous preliminary study, the investigators demonstrated significantly lower concentrations of neurofilaments in CSF of psychiatric patients compared to neurodegenerative diseases.

The main objective of this study is to validate the plasma assay of neurofilament light chain as a biomarker for the differential diagnosis of psychiatric or neurodegenerative cognitive impairment. Other biomarkers of interest (Tau, TDP-43, GFAP and UCH-L1) will also be analyzed.

A sub-part of this study will also focus on the retrospective analysis of the CSF/Plasma correlations of the different biomarkers mentioned above from tube bottom samples taken in routine care.

DETAILED DESCRIPTION:
One hundred twenty participants will be included in this study

* 30 participants suffering from psychiatric disorders (bipolar disorder or schizophrenia) without cognitive impairment
* 30 participants suffering from psychiatric disorders (bipolar disorder or schizophrenia) with cognitive impairment
* 30 participants with a biological diagnosis of Alzheimer's disease
* 30 participants with frontotemporal dementia according to Rascosky's criteria

All the participants will perform cognitive, behavioral, and psychiatric evaluation and will be have blood sample taken.

ELIGIBILITY:
Inclusion Criteria:

* haven given written consent

Participants with psychiatric conditions:

* Schizophrenia (DSM-V criteria) with or without cognitive involution
* Bipolar disorder (DSM-V criteria) with or without cognitive involution

Participants with neurodegenerative disease:

* probable or definite FTD (Rascovsky criteria 2011)
* Biological Alzheimer's disease with typical CSF (NIA-AA 2011)

Exclusion Criteria:

* Uninterviewable patient and/or missing history
* History of recent or previous head trauma with loss of consciousness
* History of ischemic or hemorrhagic stroke
* Chronic alcoholism / chronic drug use
* Progressive somatic pathology / severe metabolic disorder / poorly controlled epilepsy
* Age < 45 years
* Age > 80 years
* Electroconvulsive therapy for less than 6 months

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2028-03-22 (Estimated)

PRIMARY OUTCOMES:
neurofilament light chain | two months
  serum neurofilament light chain concentration

SECONDARY OUTCOMES:
Total tau | two months
  serum tau protein concentration
GFAP Glial fibrillary acidic protein | two months
  Serum GFAP concentration
neurofilament heavy chain (pNF-h) | two months
  Serum neurofilament heavy chain (pNF-h) concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel DOREY, MD, PHD, Principal Investigator — CH le Vinatier
Locations (2):
- France (2):
  - HCL Consultation mémoire Neurologique -Hôpital Neurologique, Bron
  - Centre Hospitalier Le Vinatier, Bron

IPD SHARING:
Plan to Share IPD: Yes
Clinical and biological IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 4 years
Access Criteria: all criterias